CLINICAL TRIAL: NCT03387540
Title: Evaluation of Reporting of Immune Checkpoint Inhibitor Associated Cardio-vascular Adverse Reactions Using International Pharmacovigilance Database
Brief Title: Evaluation of Reporting of Immune Checkpoint Inhibitor Associated Cardio-vascular Adverse Reactions
Acronym: RAFALE
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: Institute of Cardiometabolism and Nutrition, France (Other); Vanderbilt University (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, Principle investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-17-12
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Myocarditis; Cardiac Complication
Keywords: Anti-PD-1; Anti-PD-L1; Anti CTLA-4; Immune checkpoint inhibitors
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Myocarditis induced by Immune check point inhibitor: Case reported in the World Health Organization (WHO) of myocarditis of patient treated by ICI, with a chronology compatible with the drug toxicity
  Interventions: Drug: ICI

INTERVENTIONS:
Drug: ICI — Immune checkpoint inhibitor targeting either PD-1, PD-L1 or CTLA-4, and included in the following list (ATC classification): Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32).

SUMMARY:
Immune checkpoint inhibitors (ICIs) might have high grade immune-related adverse events (irAEs) on the cardio-vascular system. This study investigates reports of cardio-vascular toxicity with treatment including anti-PD1, Anti-PDL-1, and Anti CTLA4 classes using the World Health Organization (WHO) database VigiBase.

DETAILED DESCRIPTION:
ICIs have dramatically improved clinical outcomes in multiple cancer types and are increasingly being tested in earlier disease settings and used in combination. However, irAEs can occur. Here the investigators use VigiBase (http://www.vigiaccess.org/), the World Health Organization (WHO) database of individual safety case reports, to identify cases of cardiovascular adverse drug reaction following treatment with ICIs.

ELIGIBILITY:
Inclusion Criteria:

* Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017
* Adverse event reported were including the MedDRA terms: Cardiac and vascular investigations (excl enzyme tests) (HLGT), Vascular disorders (SOC), Skeletal and cardiac muscle analyses (HLT), Sudden death (PT), Sudden cardiac death (PT), Cardiac disorders (SOC), Cardiac arrhythmias (HLGT), Cardiac disorder signs and symptoms (HLGT), Cardiac neoplasms (HLGT), Cardiac valve disorders (HLGT), Congenital cardiac disorders (HLGT), Coronary artery disorders (HLGT), Endocardial disorders (HLGT), Heart failures (HLGT), Myocardial disorders (HLGT), Pericardial disorders (HLGT)
* Patients treated with ICIs included in the ATC: Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32).

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with an ICI for a cancer
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-12-02 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Cardio-vascular toxicity of ICIs. | Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017
  Identification and report of the cardio-vascular toxicity of ICIs. The research includes the report with MedDRA terms: SOC Cardiac Disorders, SOC Vascular Disorders, Sudden death (PT), Cardiac and vascular investigations (excl enzyme tests) (HLGT), Skeletal and cardiac muscle analyses (HLT). Drugs investigated are ICIs: Ipilimumab (L01XC11), Nivolumab (L01XC17), Pembrolizumab (L01XC18), Durvalumab (L01XC28), Avelumab (L01XC31), Atezolizumab (L01XC32).

SECONDARY OUTCOMES:
Causality assessment of reported cardiovascular events according to the WHO system | Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017
Description of the type of cardiotoxicity depending on the category of ICIs | Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017
Description of the duration of treatment when the toxicity happens (role of cumulative dose) | Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017
Description of the drug-drug interactions associated with adverse events | Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017
Description of the pathologies (cancer) for which the incriminated drugs have been prescribed | Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017
Description of the population of patients having a cardio-vascular adverse event | Case reported in the World Health Organization (WHO) database of individual safety case reports to 12/31/2017

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Pitié-Salpêtrière Hospital, Department of Pharmacology, CIC-1421, Pharmacovigilance Unit, INSERM., Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dressler D, Potter H. Molecular mechanisms in genetic recombination. Annu Rev Biochem. 1982;51:727-61. doi: 10.1146/annurev.bi.51.070182.003455. No abstract available. PMID 6287923
- [Result] Moslehi JJ, Salem JE, Sosman JA, Lebrun-Vignes B, Johnson DB. Increased reporting of fatal immune checkpoint inhibitor-associated myocarditis. Lancet. 2018 Mar 10;391(10124):933. doi: 10.1016/S0140-6736(18)30533-6. No abstract available. PMID 29536852
- [Result] Moslehi JJ, Salem JE, Sosman JA, Lebrun-Vignes B, Johnson DB. Reporting of immune checkpoint inhibitor-associated myocarditis - Authors' reply. Lancet. 2018 Aug 4;392(10145):384-385. doi: 10.1016/S0140-6736(18)31556-3. No abstract available. PMID 30102170
- [Result] Salem JE, Manouchehri A, Moey M, Lebrun-Vignes B, Bastarache L, Pariente A, Gobert A, Spano JP, Balko JM, Bonaca MP, Roden DM, Johnson DB, Moslehi JJ. Cardiovascular toxicities associated with immune checkpoint inhibitors: an observational, retrospective, pharmacovigilance study. Lancet Oncol. 2018 Dec;19(12):1579-1589. doi: 10.1016/S1470-2045(18)30608-9. Epub 2018 Nov 12. PMID 30442497